CLINICAL TRIAL: NCT03409523
Title: An Observational Pilot Study to Develop a Behavioral Economics Electronic Health Record Module to Guide the Care of Older Adults With Diabetes
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17-01308
Record Dates: First submitted 2017-12-26; First posted 2018-01-24 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will develop a new electronic health record module to improve guideline-compliant care of older adults with diabetes. The module will incorporate effective behavioral economics (BE) principles to improve the degree to which care of older adults is compliant with Choosing Wisely guidelines; this generally involves less aggressive targets for HbA1c, and reductions of medications other than metformin.

The implementation of the module will ultimately be triggered by medication prescribing in EPIC. The BE principles include suggesting alternatives to medications, requiring justification, setting of appropriate default order sets, and incorporation of anchoring and checklists to guide behavior. The study will involve provider workflow analysis based on observation, module user testing, and live usability testing with direct observation and semi-structure interviews.

DETAILED DESCRIPTION:
The primary objective of this study is to develop a scalable, EHR customization toolkit that applies BE insights to promote appropriate diabetes care in older adults based on the American Geriatric Society's Choosing Wisely Guideline, as to assess the acceptability of the resulting module.

ELIGIBILITY:
Inclusion Criteria:

* Providers in NYU outpatient primary care, geriatrics, or endocrine clinics at NYU who care for older adults with diabetes

Exclusion Criteria:

* None

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Providers in NYU outpatient primary care, geriatrics, or endocrine clinics at NYU who care for older adults with diabetes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Compliance with Choosing Wisely guidelines measured by number of reductions of medications | 60 Months
  The implementation of the module will ultimately be triggered by medication prescribing in EPIC.

SECONDARY OUTCOMES:
Usability measured by module user testing with direct observation and semi structured interviews | 60 Months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Troxel, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Belli HM, Chokshi SK, Hegde R, Troxel AB, Blecker S, Testa PA, Anderman J, Wong C, Mann DM. Implementation of a Behavioral Economics Electronic Health Record (BE-EHR) Module to Reduce Overtreatment of Diabetes in Older Adults. J Gen Intern Med. 2020 Nov;35(11):3254-3261. doi: 10.1007/s11606-020-06119-z. Epub 2020 Sep 3. PMID 32885374